CLINICAL TRIAL: NCT03088137
Title: Multicentre Study to Compare Efficacy and Safety of Primapur and Gonal-f in Women for Assisted Reproductive Treatment
Brief Title: Study to Compare Efficacy and Safety of Primapur and Gonal-f in Women for Assisted Reproductive Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: IVFarma LLC (Industry)
Collaborators: BridgePharm LLC (Unknown); GlobalPharma LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FSG-03-01
Record Dates: First submitted 2017-03-02; First posted 2017-03-23 (Actual); Results first posted 2019-06-06 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Infertility, Female
Keywords: in vitro fertilization
MeSH Terms: conditions — Infertility, Female | interventions — follitropin alfa

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primapur (Follitropin alfa) (Experimental)
  Interventions: Drug: Follitropin alfa (Primapur)
- Gonal-f (Follitropin alfa) (Active Comparator)
  Interventions: Drug: Follitropin alfa (Gonal-f)

INTERVENTIONS:
Drug: Follitropin alfa (Gonal-f) — Subcutaneous injection, fixed starting dose 150 IU for 5 days, maximum of 16 days of ovarian hyperstimulation
  Arms: Gonal-f (Follitropin alfa)
Drug: Follitropin alfa (Primapur) — Subcutaneous injection, fixed starting dose 150 IU for 5 days, maximum of 16 days of ovarian hyperstimulation
  Arms: Primapur (Follitropin alfa)

SUMMARY:
The purpose of this study is to show equivalence with regard to the number of oocytes retrieved between follitropin alfa (pen-injectors) Primapur® and Gonal-f® in woman undergoing IVF/ICSI

ELIGIBILITY:
Inclusion Criteria:

* Infertility due to tubal factor and/or male factor
* Age between 20 and 35 years with regular menstrual cycles of 21-35 days
* First or second cycle in the present series of ART
* BMI (body mass index) ≥ 18 ≤ 30 kg/m2
* Basal FSH (follicle stimulating hormone) < 10 IU/L (cycle day 2-5)
* E2 (estradiol) levels < 50pg/mL (cycle day 2)
* AMH (anti-mullerian hormone) ≥ 1.0 ng/ml
* Antral follicle ≥ 4 to ≤ 15 follicles (both ovaries)
* Presence of both ovaries and normal uterine cavity
* Informed consent

Exclusion Criteria:

* Presence of pregnancy
* Hypersensitivity to follitropin alfa
* Ovarian cysts
* History of ≥2 succeeding ART (assisted reproductive technology) cycles IVF (in vitro fertilization) and/or ICSI (Intracytoplasmic sperm injection) before the study cycle
* Previous history of severe ovarian hyperstimulation syndrome
* Presence of polycystic ovaries (PCO)
* Presence of endometriosis and hydrosalpinx
* Presence of uterine disorders
* History of poor (< 4 oocytes) or hyper (> 25 oocytes) responses to FSH treatment at dose 150 IU and GnRH-antagonist (gonadotropin-releasing hormone) protocol
* Premature ovarian failure
* Ectopic pregnancy (3 month before the study cycle)
* Presence of clinically significant systemic disease
* Presence of chronic cardiovascular, hepatic, renal or pulmonary disease
* Presence of endocrine disorder
* Neoplasia
* Male infertility without mobile spermatozoa in the ejaculate, that need MESA (Microsurgical epididymal sperm aspiration)/TESE (testicular sperm extraction)/TESA (testicular sperm aspiration)
* Smoking > 10 cigarettes/day
* Narcomania, alcoholism
* Planned PGS (preimplantation genetic screeneing) /PGD (preimplantation genetic diagnosis)

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2017-02-08 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - AltraVita IVF clinic, Moscow
  - Perinatal Medical Center, Moscow
  - Clinical Hospital Lapino, Moscow Oblast

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] M. Polzikov, Z. Barakhoeva, S. Yakovenko, M. Ovchinnikova, L.Vovk, Y. Fetisova. A multicenter, randomized study comparing the efficacy of follitropin alpha biosimilar and the original follitropin alpha. Abstracts of the 35th Annual Meeting of the ESHRE, Vienna, Austria 24 to 26 June 2019 (abstract P-649), Human Reproduction, 2019; Vol. 34, Suppl. 1, p. i439.
- [Result] Barakhoeva Z, Vovk L, Fetisova Y, Marilova N, Ovchinnikova M, Tischenko M, Scherbatyuk Y, Kolotovkina A, Miskun A, Kasyanova G, Teterina T, Zorina I, Belousova N, Morozova E, Yakovenko S, Apryshko V, Sichinava L, Shalinsmall a, Cyrillic R, Polzikov M. A multicenter, randomized, phase III study comparing the efficacy and safety of follitropin alpha biosimilar and the original follitropin alpha. Eur J Obstet Gynecol Reprod Biol. 2019 Oct;241:6-12. doi: 10.1016/j.ejogrb.2019.07.032. Epub 2019 Jul 26. PMID 31400644
- [Result] Barakhoeva Z.B., Vovk L.A., Zorina I.V., Belousova N.Y., Teterina T.A., Yakovenko S.A., Apryshko V.P., Fetisova Y.A., Marilova N.A., Morozova E.G., Ovchinnikova M.M., Tishenko M.A., Sherbatyuk Y.V., Kolotovkina A.V., Miskun A.A., Kasyanova G.V., Sichinava L.G., Shalinа R.I., Polzikov M.A. Major results of a phase III comparative multicenter study on the follitropin alfa biosimilar (Primapur®) and the original follitropin alfa (Gonal-f®). Akusherstvo, ginekologiya i reprodukciya. 2018;12(3):5-16. (In Russ.) https://doi.org/10.17749/2313-7347.2018.12.3.005-016
- [Derived] Polzikov M, Blinov D, Barakhoeva Z, Vovk L, Fetisova Y, Ovchinnikova M, Tischenko M, Zorina I, Yurasov V, Ushakova T, Sergeyev O. Association of the Serum Folate and Total Calcium and Magnesium Levels Before Ovarian Stimulation With Outcomes of Fresh In Vitro Fertilization Cycles in Normogonadotropic Women. Front Endocrinol (Lausanne). 2022 Feb 11;13:732731. doi: 10.3389/fendo.2022.732731. eCollection 2022. PMID 35222266
- See also: European Journal of Obstetrics & Gynecology and Reproductive Biology Volume 241, October 2019, Pages 6-12 — https://doi.org/10.1016/j.ejogrb.2019.07.032

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at 3 In Vitro Fertilisation (IVF) centers in Russian Federation from 08.02.2017 - 17.08.2018.
Pre-assignment Details: Of 118 participants: 8 were reported as screening failures prior the group assignment.
Groups:
- Primapur (Follitropin Alfa): Follitropin alfa (Primapur): Subcutaneous injection (pen-injector), fixed starting dose 150 IU for 5 days, maximum of 16 days of ovarian hyperstimulation
- Gonal-f (Follitropin Alfa): Follitropin alfa (Gonal-f): Subcutaneous injection (pen-injector), fixed starting dose 150 IU for 5 days, maximum of 16 days of ovarian hyperstimulation
Period: Overall Study
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Started | 55 | 55
Completed | 55 | 55
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa) | Total
Number analyzed (Participants) | 55 | 55 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] — Mean (Standard Deviation)
  years | 31.3 (2.68) | 30.0 (2.71) | 30.65 (2.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 55 | 110
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 55 | 55 | 110
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Russia | 55 | 55 | 110
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] — kg/m2
  kg/m2 | 22.0 (2.69) | 22.3 (3.06) | 22.15 (2.87)
Duration of infertility [Mean (Standard Deviation); unit: month] — month
  month | 46.4 (32.4) | 36.9 (26.6) | 41.65 (28.22)
Antral follicle [Mean (Standard Deviation); unit: Number of antral follicles] — Mean (Standard Deviation)
  Number of antral follicles | 11.2 (3.2) | 12.4 (2.4) | 11.80 (2.87)
Anti-mullerian hormone (AMH) [Mean (Standard Deviation); unit: ng per ml] — Mean (Standard deviation)
  ng per ml | 4.57 (2.96) | 5.47 (3.82) | 5.02 (3.43)
Follicle stimulating hormone (FSH) [Mean (Standard Deviation); unit: IU/l] — IU per l
  IU/l | 6.46 (1.86) | 6.76 (1.89) | 6.61 (1.87)
Estradiol [Mean (Standard Deviation); unit: pg/ml] | 35.87 (12.67) | 33.82 (12.45) | 34.85 (12.54)
Cause of infertility [Count of Participants; unit: Participants] — Patients with the determined cause of infertility
  Participants
    Tubal factor | 21 | 18 | 39
    Male factor | 21 | 27 | 48
    Tubal and male factors | 13 | 10 | 23

OUTCOME MEASURES:

1. Primary Outcome: Oocytes (Intention-to-Treat, ITT)
Description: The total number of retrieved oocytes at the day of ovum pick-up. No more than 37 hours from the introduction of the trigger of ovulation (hCG or GnRH-agonist). The equivalence in the number of retrieved oocytes was tested using a predetermined equivalence margin of +/- 3.4 oocytes.
Time Frame: From date of randomization up to 18 days
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: Number of retrieved oocytes
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Number of retrieved oocytes | 12.16 (7.28) | 11.62 (6.29)
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Equivalence — Study power of at least 80% at a significance level (alpha error) 5% and a pre-determined clinical equivalence margin of +/- 3.4 oocytes for the relevant population; p = 0.002, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.546, 95% CI 2-sided [-2.026 to 3.116], Standard Deviation 1.297

2. Secondary Outcome: Number of Follicles With Size ≥ 16 mm
Description: The number of follicles 16 mm or over in diameter at the day of hCG (or GnRH-agonist) administration
Time Frame: From date of randomization up to 16 days
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: Number of follicles
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Number of follicles | 12.09 (6.159) | 11.38 (4.965)
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Superiority; p = 0.806, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.709, 95% CI 2-sided [-1.405 to 2.824], Standard Deviation 1.067

3. Secondary Outcome: Mature Oocytes
Description: The number of mature oocytes (MII stage of development)
Time Frame: From date of randomization up to 18 days
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: Number of mature oocytes (MII stage)
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Number of mature oocytes (MII stage) | 9.64 (6.270) | 9.86 (5.546)
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Superiority; p = 0.617, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.218, 95% CI 2-sided [-2.455 to 2.019], Standard Deviation 1.129

4. Secondary Outcome: Fertilised Oocytes
Description: The number of fertilised oocytes with the presence of two pronuclei: 2PN
Time Frame: From date of randomization up to 19 days
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: Number of oocytes with 2PN
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Number of oocytes with 2PN | 8.127 (6.608) | 8.764 (5.850)
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Superiority; p = 0.445, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.636, 95% CI 2-sided [-2.995 to 1.723], Standard Deviation 1.190

5. Secondary Outcome: Percentage of Patients With Embryo Transfer
Description: The number of patients (and percentage) with embryo transfers on days 3 and 5 after ovum pick-up
Time Frame: From date of randomization up to 25 days
Population: Per Protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 49 | 49
Participants
  Embryo transfer on day 3 (%) | 11 | 9
  Embryo transfer on day 5 (%) | 38 | 40
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Superiority; p = 0.623, ANOVA

6. Secondary Outcome: Total Dose of Follitropin Alfa
Description: The total dose of the follitropin alfa administrated during the ovarian hyperstimulation protocol (measured in International Units - IU)
Time Frame: From date of randomization up to 16 days
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: Total dose (IU)
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Total dose (IU) | 1532.7 (267.2) | 1517.9 (255.2)
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Superiority; p = 0.488, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 14.9, 95% CI 2-sided [-83.9 to 113.6], Standard Deviation 49.8

7. Secondary Outcome: Number of Days of Follitropin Alfa Treatment
Description: The duration of ovarian hyperstimulation protocol (at the day of trigger of ovulation)
Time Frame: From date of randomization up to 16 days
Population: Intention-to-Treat
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Days | 9.745 (1.075) | 9.727 (1.027)
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Superiority; p = 0.629, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.018, 95% CI 2-sided [-0.379 to 0.416], Standard Deviation 0.201

8. Secondary Outcome: Number of Patients With Follitropin Alfa Dose Correction
Description: The number of dose adjustments during the ovarian hyperstimulation protocol (increment 25-50 IU)
Time Frame: From date of randomization up to 16 days
Population: Intention-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Participants | 13 | 11
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); Test type: Superiority; p = 0.644, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Number of Patients With Cycle Cancellation
Description: The number of the ovarian hyperstimulation protocol cancellation (at the day of trigger of ovulation)
Time Frame: From date of randomization up to 16 days
Population: Intention-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Participants | 0 | 0

10. Secondary Outcome: Number of No-responders
Description: The number of patients with no response to follitropin alfa treatment (absence of growing follicles, no any oocytes obtained at the day of ovum pick-up)
Time Frame: From date of randomization up to 8 days
Population: Intention-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 55 | 55
Participants | 0 | 0

11. Secondary Outcome: Percentage of Patients With Serum hCG More Than 25 IU/l
Description: Biochemical pregnancy test: serum hCG more than 25 IU/l (days 12-17 after embryo transfer)
Time Frame: From date of randomization up to 42 days
Population: Per Protocol
Measure: Number (95% Confidence Interval); unit: Percentage of patients (%)
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 49 | 49
Percentage of patients (%) | 34.7 [21.4 to 48.0] | 36.7 [23.2 to 50.2]
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); 95% confidence intervals (CIs) of point estimates were calculated using the exact binomial distribution (Clopper-Pearson method) for proportions; Test type: Superiority; p = 0.833, Chi-squared; Mean Difference (Final Values) = -2.0, 95% CI 2-sided [-21.0 to 17.0]

12. Secondary Outcome: Percentage of Patients With the Evidence for Clinical Pregnancy
Description: Confirmation of clinical pregnancy: ultrasound detection of intrauterine gestational sac and heart activity
Time Frame: The 10th week after embryo transfer
Population: Per Protocol
Measure: Number (95% Confidence Interval); unit: Percentage of patients (%)
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
Number analyzed (Participants) | 49 | 49
Percentage of patients (%) | 26.5 [14.1 to 38.9] | 32.7 [19.6 to 45.8]
Statistical Analysis 1: Comparison: Primapur (Follitropin Alfa) vs Gonal-f (Follitropin Alfa); [analysis description as in outcome 11, analysis 1]; Test type: Superiority; p = 0.507, Chi-squared; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-24.3 to 11.9]

ADVERSE EVENTS:
Time Frame: 1 year, 6 month
Arm/Group | Primapur (Follitropin Alfa) | Gonal-f (Follitropin Alfa)
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/55 | 2/55
Other Adverse Events (participants affected / at risk) | 21/55 | 13/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primapur (Follitropin Alfa) (N=55) | Gonal-f (Follitropin Alfa) (N=55)
Ovarian hyperstymulation syndrome (Reproductive system and breast disorders) | 0 (0) | 2 (2) — Patients with positive pregnancy test
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — iatrogenic bladder injury during transvaginal ovarian puncturing
Threatened miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Primapur (Follitropin Alfa) (N=55) | Gonal-f (Follitropin Alfa) (N=55)
Spontaneous miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Early Toxicosis During Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abnormal vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Menses (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian hyperstimulation syndrome (Reproductive system and breast disorders) | 4 (4) | 2 (2) — Patients with negative pregnancy test
Decrease in breast sensitivity (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Spotting (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Lower abdominal pain (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 4 (4)
Lower abdominal pain (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Pains in the lower abdomen (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Laboratory investigations (Investigations) | 1 (1) | 0 (0) — Erythrocyte level increase in urine
Sternum pain (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Drowsiness (Nervous system disorders) | 1 (1) | 0 (0)
Fatigue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abnormal vaginal bleeding (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Spotting (Reproductive system and breast disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT03088137/Prot_SAP_000.pdf